CLINICAL TRIAL: NCT04893174
Title: A Phase 1, Open Label, Dose Escalation Study to Evaluate the Safety and Tolerability After Intra Articular (IA) Injection of UMC119-06-05 in Adult Subjects With Mild to Moderate Knee Osteoarthritis(KOA).
Brief Title: Mesenchymal Stem Cells for The Treatment of Knee Osteoarthritis (KOA).
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meridigen Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UMC119-06-05-KOA-01
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2022-12

CONDITIONS: Osteoarthritis, Knee
Keywords: KOA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Cohort 1 : Low does UMC119-06-05 + Hyaluronic acid； Cohort 2 : High does UMC119-06-05 + Hyaluronic acid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- UMC119-06-05 (Experimental): Human Umbilical Cord Derived-Mesenchymal Stem Cells. Subjects will receive a single-dose intra-articular (IA) injection of UMC119-06-05 followed by an IA injection of hyaluronic acid.
  Interventions: Biological: UMC119-06-05; Device: Hyaluronic acid

INTERVENTIONS:
Biological: UMC119-06-05 — Subjects will receive a single-dose IA injection of UMC119-06-05 followed by an IA injection of hyaluronic acid.
  Cohort 1: Low does UMC119-06-05 Cohort 2: High does UMC119-06-05
Device: Hyaluronic acid — IA injection of hyaluronic acid.

SUMMARY:
The clinical study with UMC119-06-05 is designed to investigate the safety in patients with mild to moderate knee osteoarthritis (KOA). This will be a dose escalation, open label, single-center study in adult with mild to moderate knee osteoarthritis. UMC119-06-05 is ex vivo cultured human umbilical cord tissue-derived mesenchymal stem cells product which is intended for treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA), also known as degenerative joint disease, is the most common type of arthritis diagnosed. KOA is typically the result of wear and tear and progressive loss of articular cartilage. The prevalence of the Knee osteoarthritis will continue to increase as life expectancy and obesity rises. Osteoarthritis is typically a progressive disease that may eventually lead to disability. The intensity of the clinical symptoms may vary from each individual. However, they typically become more severe, more frequent, and more debilitating over time.The intensity of the clinical symptoms may vary from each individual. However, they typically become more severe, more frequent, and more debilitating over time.

The rate of progression also varies for each individual. Common clinical symptoms include knee pain that is gradual in onset and worse with activity, knee stiffness and swelling, pain after prolonged sitting or resting, and pain that worsens over time. Treatment for knee osteoarthritis begins with conservative methods and progresses to surgical treatment options when conservative treatment fails. While medications can help slow the progression of RA and other inflammatory conditions, no proven disease-modifying agents for the treatment of knee osteoarthritis currently exist. Among the more innovative, experimental therapies, mesenchymal stromal cells (MSCs) are proposed as a novel therapy with potential in treatment of KOA.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory subjects with osteoarthritis of the knee with symptoms for at least 3 months, that may be taking conservative therapy (e.g. oral anti-inflammatory medication), and/or undergoing physical therapy. In subjects with bilateral knee osteoarthritis, the more symptomatic knee will be the target knee.
2. Subjects of age between ≥40 through ≦ 90 years.
3. Subject diagnosed with knee osteoarthritis of grade II and III according to the Kellgren-Lawrence Grading Scale on the target knee.
4. Subject with joint pain equal or greater than 7 (total pain score 24 point) on the target knee assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).
5. Subject or legal guardian is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided, and has had the opportunity to discuss the study with the investigator or designee.
6. Women of child-bearing potential should have a negative urine pregnancy test prior to administration of investigational product, and the subject must agree within at least 4 weeks after the study administration to use a double barrier method of birth control.UNLESS they meet the following criteria:(1) Post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum Follicle Stimulating Hormone (FSH) levels > 40mIU/mL, OR; (2) 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy.
7. If a male and heterosexually active with a female of childbearing potential, the subject must agree within at least 4 weeks after the study administration to use a double barrier method of birth control (or must have been surgically sterilized) and to not donate sperm.

Exclusion Criteria:

1. Subjects with body mass index (BMI) over 40.
2. Subjects with knee deformity (knee varus or valgus greater than 10 degrees) on the target knee.
3. Subjects with acute inflammation or tense effusion (e.g., infection), or bleeding on the target knee as judged by principal investigator (PI).
4. Subjects with ligament instability (cruciate ligaments or collateral ligaments) or ligament laxity of the target knee as judged by PI.
5. Subjects with a history of surgery of articular injury, ligament reconstruction and meniscus repair on the target knee joint within previous 6 months.
6. Subjects with history of arthroscopic surgery in the target knee in the past 6 months or planned to have arthroscopy surgery during the trial period (e.g., scheduled for/awaiting arthroscopy or a knee replacement procedure)
7. Subjects with history of knee replacement procedure on the target knee.
8. Subjects with intra-articular infiltration of any treatments on the target knee (such as hyaluronic acid, corticosteroids or platelet rich plasma (PRP)) in the last 3 months prior to study inclusion.
9. Subjects with known history of osteoarthritis of hip or ankle.
10. Subjects with known history of any systemic autoimmune rheumatic disease including but not limited to: Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, lymphoma, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis.
11. Subjects with Rheumatoid Factor levels (>15.9 IU/mL) in laboratory tests.
12. Subjects with joint diseases (except knee osteoarthritis) or infectious arthritis on the target knee considered by investigator not eligible to enter the study.
13. Subjects who are known to be infected with HIV.
14. Subjects with active hepatitis B or active hepatitis C.
15. Subjects who have a significant concomitant illness as judged by principal investigator (PI) including, but not limited to:

    1. Severe renal insufficiency (eGFR < 30 mL/min/1.73 m2); or
    2. hepatic (e.g. Child-Pugh Class C); or
    3. Severe congestive heart failure (NYHA class 3 and 4); or
    4. Severe pulmonary dysfunction, including severe chronic obstructive pulmonary disease (COPD) and history of lung resection; or
    5. Any type of malignancy; or
    6. Uncontrolled Diabetes Mellitus (HbA1c > 10%)
16. Subjects with uncorrected hematology test including, but not limited to:

    1. Hemoglobin < 8 g/dl; or
    2. White blood cell count < 3,000/mm3; or
    3. International normalized ratio (INR) of Coagulopathy >1.5; or
    4. Platelet count < 80,000/mm3
17. Subjects who have the following conditions in laboratory tests:

    1. >2 × upper limit of normal for alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ; or
    2. Total bilirubin > 1.5 mg/dl
18. Subjects with known history of allergy or hypersensitivity to any component of investigational product, including dimethyl sulfoxide, cell therapies, or hyaluronic acid.
19. Subjects with known history of allergy or hypersensitivity to any concomitant medications, or rescue medications.
20. Subjects who have a significant skin disease at the injection site on target knee as judged by principal investigator (PI).
21. Subjects who are pregnant (or planning to become pregnant within 2 years of investigational product treatment) or lactating.
22. Participation in another clinical trial or treatment (e.g., immunosuppressant therapies, systemic steroids, cytotoxic drugs, chemotherapy, radiation therapy, new investigational drugs or cell therapy) within 3 months prior to inclusion in the study.
23. Contraindication to MRI:

    * Indwelling medical devices such as pacemakers, aneurysm clip, etc.
    * Indwelling metal from any other cause (trauma, etc.). To be excluded with history and/or radiographs, as necessary
24. Other pathologic conditions or circumstances that difficult participation in the study according to medical criteria.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The incidence and frequency of adverse events related to administration of UMC119-06-05. | 1 months from the day of administration
  Incidence of Treatment-Emergent Adverse Events (TEAEs). Incidence of withdrawals due to Adverse Events(AEs).

SECONDARY OUTCOMES:
Changes of total score in the Western Ontario and McMaster (WOMAC) assessment on the target knee. | from baseline up to 52 weeks after administration
  Improvement in total score (pain subscale, and stiffness subscale, and physical function subscale) as assessed by mean change in WOMAC index.
Changes of arthritis pain on target knee using the 100-mm visual-analogue scale (VAS). | from baseline up to 52 weeks after administration
  VAS scale range 0 to 100 mm, with higher scores indicates greater pain intensity. A decrease in score represents a decrease in disease related pain of knee.
Whole Organ Magnetic Resonance Imaging Score (WORMS). | from baseline up to 52 weeks after administration
  Changes on the target knee for knee cartilage and the joint soft tissues assessed by Whole Organ Magnetic Resonance Imaging Score (WORMS) using magnetic resonance imaging (MRI) of T2 mapping.
Changes in Kellgren-Lawrence (K-L) grading and joint space on target knee. | from baseline up to 52 weeks after administration
  The severity of knee OA was defined as kellgren-lawrence (K-L) classification criteria. Changes from baseline to post-treatment visits on the target knee for Kellgren-Lawrence (K-L) grading and joint space in X-ray examination results.
Amount of rescue medications required. | at first 4 weeks, first 28 weeks and the whole study period.
  Total amount of acetaminophen or non-steroidal anti-inflammatory drugs (NSAID)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No